# Golimumab effect in the modulation of gut microbiota in Ulcerative Colitis. Pilot Study.

**Protocol Code:** GOLI2015 v1 10/11/2015

**Promotor:** Merck & Co., Inc.

Financing: This project will be funded by Merck & Co., Inc

Investigador principal: Dr. Xavier Aldeguer Manté, Head of Gastroenterology Service,

Hospital Universitari de Girona, Dr. Josep Trueta.

# Centers where the study will take place:

Hospital Universitari de Girona, Dr. Josep Trueta Av de França S/N, 17007, Girona, Spain

Hospital de Santa Caterina

Carrer del Dr. Castany, s/n, 17190 Salt, Girona, Spain

Collaborating centers: Centers of Catalonia, that will wish to participate after the

approval of this project

**Duration:** 26 months, Starts in May 2016

## 1. BACKGROUND

Recently, a consistent body of evidence indicates that the gut microbiota ability to modulate and direct the host immune response is considered one of the pivotal factors that modulate the delicate balance between health and disease in digestive diseases (1). In the case of inflammatory bowel disease (IBD), the gut microbiota has a central role in maintaining the microbiological homeostasis of the patient (2, 3). Recent studies describe the existence of different patterns of intestinal microbiota from patients with IBD and healthy individuals (4, 5). The alteration of the microbiological pattern not associated with disease is known as dysbiosis and is directly related to the degree of inflammation of the intestinal mucosa, and, thus, the clinic status: a greater dysbiosis, greater clinical correlation with disease state, so that the gut microbiota is a direct marker of the state of colonic inflammation (6).

The state of dysbiosis is measured through different microbiological indices of the total population of bacteria in the colon. Changes in rates of these indices are the parameters that are measured to characterize the gut microbiota of the patients. In the case of ulcerative colitis (UC) studies have shown that intestinal microbiota is a central factor in maintaining the balance between deep remission and the presence of a flare-up (7, 8). Despite advances, in-depth knowledge of how the gut microbiota interacts with the intestinal mucosa and alters the intestinal barrier and the molecular/genetic mechanism is still unknown. Some genes and associated cofactors have been identified but the exact mechanism of interaction has not yet been described. The data indicate that, presumably, the mechanism of regulation is a multifactorial process (9, 10).

In this way, a deep understanding of gut microbiota and its interactions with the host and the colon will be of great interest, in order to shape the future of IBD treatment, especially of UC. Thus, IBD patients' intestinal microbiota could be either a therapeutic target itself (fecal transplantation) or be consider as an adjustable adjuvant with immunomodulators (11, 12).

The group of anti-TNF $\alpha$  drugs are the most recently incorporated in the therapeutic arsenal of UC, in some cases changing the natural curse of the disease. However, it is still unknown how these drugs modulate the intestinal microbiota and how they interfere with it, although, probably,

they develop a role. Recent results from studies by our group, indicate that on entering clinical remission, gut microbiota is modified to patterns less related with dysbiosis (13, 14,15, 16). Given the increasing importance of the use of anti-TNF $\alpha$  drugs, it is of great interest to discriminate between the patterns associated with dysbiosis and those related with healthy mucosa, and how they are modified as a result of the use of anti-TNF $\alpha$  drugs. In this way, previous results of our group analyzing the changes of intestinal microbiota associated with Adalimumab anti-TNF $\alpha$  drug treatment have shown that during the progression of the patient into remission, the mucosal dysbiosis pattern changes (17). On the other hand, our group has also observed that after drug treatment failure, the gut microbiota returns to a pattern closer to dysbiosis. For that reason, gut microbiota could be considered as an excellent indicator of the real drug effectiveness in the patient.

Regarding Golimumab, a recently introduced anti-TNF $\alpha$  drug therapy in UC, it is still unknown how it is able to modulate the intestinal microbiota to remission-related patterns, since to date there are not available studies about the relationship between Golimumab and this phenomenon.

The use of prebiotics and probiotics has shown some effectiveness as adjuvants in the treatment of UC (18). For that reason, further characterization of the gut microbiota patterns is very important to develop new strategies for adjuvant ability to modulate it, especially in patients receiving anti-TNF $\alpha$  drugs and do not achieve complete remission. Similarly to recent studies, we suggest that the modulation of gut microbiota could optimize the response outcomes in patients treated with Golimumab.

In conclusion, based on current trends in the literature, we suggest that modulation of the intestinal microbiota and the characterization of remission-related patterns, will have a huge impact on the management of patients with UC. Moreover, the modulation of gut microbiota together with the anti-TNF $\alpha$  drug effectiveness could be the most promising field in the management of inflammatory bowel disease.

#### 2. HYPOTHESIS AND OBJECTIVES

#### 2.1 Hypothesis

- 1. Intestinal microbiota profile change according UC activity.
- 2. The Intestinal microbiota profile correlated to clinical remission is represented by stable intestinal microbiota biodiversity.
- 3. Determination of Intestinal Microbiota is a useful tool to measure Golimimab efectiveness in patients naïve to anti-TNF treatment and patients recurrent to anti-TNF treatment.

# 2.2 Objectives

- To correlate clinical remission under Golimumab treatment with stable intestinal microbiota profile biodiversity
- 2. To characterize the pattern of intestinal microbiota associated with the use of Golimumab and temporal dynamics of microbial change.
- Assess the effect of golimumab on the degree of colic dysbiosis in the treatment of CU naive to Golimumab.

#### 3. MATERIAL AND METHODS

## 3.1 Type of study/design

Multicentrer transversal pilot Study

# 3.2 Study population

The proposed study will include 15 UC anti-TNF $\alpha$  naïve patients from Hospital Universitari Dr. Josep Trueta, Hospital Santa Caterina and Hospitals collaborators. We will consider remission when patients have an endoscopic Mayo score  $\leq 1$ , and activity index score, Mayo= 0 points.

## 3.2.1 Inclusion criteria

- > 18 years
- Signed the informed consent
- Anti-TNFα naïve
- Screening for opportunistic infections

#### 3.2.2 Exclusion criteria

- Active tuberculosis or another chronic infections
- Antibiotic treatment prior 1 month
- Probiotics & Prebiotics
- Gestation and lactation
- Heart disfunction
- Colectomy

## 3.3 Interventions

#### 3.3.1 Treatments

GOLIMUMAB induction with 200mg at week 0, and 100mg at week 2. Under 70kg, the follow up treatment will be 50mg/month, and 100mg/month in patients over 70kg, as clinical practice.

#### 3.4 Variables

## 3.4.1 Demographic variables

- **Age** expressed in years (y)
- Sex Male (M)/ Female (F)
- Weight expressed in IMC
- Ethnic: Caucasian/ African/ Asiatic/ American
- Tobacco: YES / NO / EX-Smoker
- Age of UC diagnosis expressed in years (y)
- Familiar Antecedents (YES/NO) which kind of disease?
- Localization Left (L)/ Righ (R) / extended (E)

#### 3.4.2 Clinical variables

- **Mayo clinic score** (Clinical colitis activity index) (Schroeder KW *et al. NEngl J Med* 1987; 317: 1625–9). Score range: 0-9 points

- CRP (C-reactive protein): blood C-reactive protein concentration (mg/L)
- **Faecal calprotectin**: stool sample expressed in concentration of calprotectin in ug for g of feces (ug/g)

# -Standard Analysis:

**Hemoglobin**: blood hemoglobin concentration (g / dl) **Platelets**: blood platelets concentration (x10<sup>3</sup>/ ul) **Leucocytes**: blood leucocytes concentration (x10<sup>3</sup>/ ul)

**Albumin**: blood albumin concentration (g / dl)

Creatinine levels: blood creatinine concentration (mg/ dl)

#### 3.4.3 Endoscopic variables

Mayo (Endoscopic score of Ulcerative Colitis) (Schroeder KW et al. 1987).
Mayo Endoscopic Score is based only on Endoscopic Findings. Mayo Score range from 0 to 3.

**Note:** We will send the image in a centralization digital platform, where we will reevaluate the Mayo score with 2 independent professionals, in order to have an objective score.

## 3.4.4 Microbiological variables

- Operational Taxonomic Units (OTUs)
- Abundance and bacterial load.

#### 3.5 Methods

The proposed study will include 15 UC patients over 18 years, that have signed the informed consent, subjected to treatment with anti-TNF $\alpha$  by clinical practice and who have made screening for opportunistic infections. Patients will be anti-TNF $\alpha$  naïve patients.

Stool samples will be collected before starting Anti-TNF treatment (M0), and then every 3 months (M1, M2, M3 and M4) to complete the study. The monitoring period shall be one year. We will be also collected at M0, M1, M2, M3 & M4 demographic variables (age, sex, tobacco, age of diagnosis, localization,...), clinical data (Mayo clinical score, CRP, albumin, hemoglobin, creatinine, leucocytes, platelets...), microbiological variables, also a 4 calprotectin determinations (at baseline, at week12, at 6 months and at the end of the study as a clinical practice) and Mayo endoscopic index (at baseline and at the end of the monitoring period as a clinical practice). Follow-up visits will also take place within routine clinical practice. For better follow-up the evolution of the patient we propose an additional test as a clinical practice, but optional, a rectosigmoidoscopy at week 12 after starting Anti-TNF treatment.

We will consider remission when patients have an endoscopic Mayo score ≤1, and activity index score, Mayo clinical score =0 points.

Moreover, depending on the evolution of the patient, additional tests shall also be performed as routine clinical protocol during the monitoring period.

#### 3.5.1 Sample processing

#### **DNA Extraction:**

Before microbiological analyses, genomic DNA of 16s RNA gene will be extracted using NucleoSpin® Soil Kit (Machery-Nagel GmbH & Co., Germany). DNA concentration will be determined with Qubit® BR (Invitrogen) Kit.

## Bacterial 16S rRNA Gene Amplification by Pyrosequencing

#### Sequence Editing and Analysis

High-quality consensus sequences were obtained and manually refined with the Bioedit software package. Alignments were carried out with ClustalW24 software. Consensus sequences were compared with those in GenBank and the Ribosomal Database Project by using BLASTN 2.2.10. Sequences were grouped by number of operational taxonomic units or phylotypes with the DOTUR program26 using the farthest neighbor method at a precision level of 0.01, i.e., 99% minimum similarity for any pair of sequences to belong to the same phylotype, on a distance matrix with the Jukes-Cantor correction calculated with the DNADIST program of the Phylip software package.

## 3.6 Statistical analysis

Statistical analysis was performed with the SPSSx version 11.0. Significance of distances between groups was checked using an analysis of variance. Pearson\_s x2 test was used to compare the prevalence of genus and species.

Clinical and laboratory data will be correlated with the values of quantitative microbial indices using Receiver Operating Characteristic (ROC) curves.

# 4. BIBLIOGRAPHY

- 1. Geuking MB, Köller Y, Rupp S, McCoy KD. The interplay between the gut microbiota and the immune system. Gut Microbes. 2014 May-Jun;5(3):411-8.
- 2. Sartor RB. Microbial influences in inflammatory bowel diseases. Gastroenterology. 2008 Feb;134(2):577-94.
- 3. Asquith M, Powrie F. An innately dangerous balancing act: intestinal homeostasis, inflammation, and colitis-associated cancer. J Exp Med. 2010 Aug 2;207(8):1573-7.
- 4. Manichanh C, Rigottier-Gois L, Bonnaud E, Gloux K, Pelletier E, Frangeul L, Nalin R, Jarrin C, Chardon P, Marteau P, Roca J, Dore J. Reduced diversity of faecal microbiota in Crohn's disease revealed by a metagenomic approach. Gut. 2006 Feb;55(2):205-11. Epub 2005 Sep 27.
- 5. Walujkar SA, Dhotre DP, Marathe NP, Lawate PS, Bharadwaj RS, Shouche YS. Characterization of bacterial community shift in human Ulcerative Colitis patients revealed by Illumina based 16S rRNA gene amplicon sequencing. Gut Pathog. 2014 Jun 14;6:22.
- 6. Walker AW, Sanderson JD, Churcher C, Parkes GC, Hudspith BN, Rayment N, Brostoff J, Parkhill J, Dougan G, Petrovska L. High-throughput clone library analysis of the mucosa-associated microbiota reveals dysbiosis and differences between inflamed and

- non-inflamed regions of the intestine in inflammatory bowel disease. BMC Microbiol. 2011 Jan 10;11:7.
- 7. Vigsnaes LK, van den Abbeele P, Sulek K, Frandsen HL, Steenholdt C, Brynskov J, Vermeiren J, van de Wiele T, Licht TR. Microbiotas from UC patients display altered metabolism and reduced ability of LAB to colonize mucus. Sci Rep. 2013;3:1110.
- 8. Varela E, Manichanh C, Gallart M, Torrejón A, Borruel N, Casellas F, Guarner F, Antolin M. Colonisation by Faecalibacterium prausnitzii and maintenance of clinical remission in patients with ulcerative colitis. Aliment Pharmacol Ther. 2013 Jul;38(2):151-61.
- 9. Maccaferri S, Biagi E, Brigidi P. Metagenomics: key to human gut microbiota. Dig Dis. 2011;29(6):525-30.
- 10. McHardy IH, Goudarzi M, Tong M, Ruegger PM, Schwager E, Weger JR, Graeber TG, Sonnenburg JL, Horvath S, Huttenhower C, McGovern DP, Fornace AJ Jr, Borneman J, Braun J. Integrative analysis of the microbiome and metabolome of the human intestinal mucosal surface reveals exquisite inter-relationships. Microbiome. 2013 Jun 5;1(1):17.
- 11. Allegretti JR, Hamilton MJ. Restoring the gut microbiome for the treatment of inflammatory bowel diseases. World J Gastroenterol. 2014 Apr 7;20(13):3468-74.
- 12. Lee KN, Lee OY. Intestinal microbiota in pathophysiology and management of irritable bowel syndrome. World J Gastroenterol. 2014 Jul 21;20(27):8886-97.
- 13. Martinez-Medina M, Aldeguer X, Gonzalez-Huix F, Acero D, Garcia-Gil LJ. Abnormal microbiota composition in the ileocolonic mucosa of Crohn's disease patients as revealed by polymerase chain reaction-denaturing gradient gel electrophoresis. Inflamm Bowel Dis. 2006 Dec;12(12):1136-45.
- Lopez-Siles M, Martinez-Medina M, Busquets D, Sabat-Mir M, Duncan SH, Flint HJ, Aldeguer X, Garcia-Gil LJ. Mucosa-associated Faecalibacterium prausnitzii and Escherichia coli co-abundance can distinguish Irritable Bowel Syndrome and Inflammatory Bowel Disease phenotypes. Int J Med Microbiol. 2014 May;304(3-4):464-75.
- Lopez-Siles M, Martinez-Medina M, Abellà C, Busquets D, Sabat-Mir M, Duncan SH, Aldeguer X, Flint HJ, Garcia-Gil LJ. Mucosa-associated Faecalibacterium prausnitzii phylotype richness is reduced in inflammatory bowel disease patients. Appl Environ Microbiol. 2015 Aug 21. PubMed PMID: 26296733.
- 16. Lopez-Siles M, Martinez-Medina M, Surís-Valls R, **Aldeguer X**, Sabat-Mir M, Duncan SH, Flint HJ, Garcia-Gil LJ. Changes in the Abundance of Faecalibacterium prausnitzii Phylogroups I and II in the Intestinal Mucosa of Inflammatory Bowel Disease and Patients with Colorectal Cancer. Inflamm Bowel Dis. 2016 Jan;22(1):28-41.
- 17. Busquets D, Mas-de-Xaxars T, López-Siles M, Martínez-Medina M, Bahí A, Sàbat M, Louvriex R, Miquel-Cusachs JO, Garcia-Gil JL, **Aldeguer X**. Anti-tumour Necrosis Factor Treatment with Adalimumab Induces Changes in the Microbiota of Crohn's Disease. J Crohns Colitis. 2015 Jul 4. PubMed PMID: 26142465.
- 18. Verbeke KA, Boesmans L, Boets E. Modulating the microbiota in inflammatory bowel diseases: prebiotics, probiotics or faecal transplantation? Proc Nutr Soc. 2014 Nov;73(4):490-7.

# **BUDGET**

| MATERIAL | |
|-------------------------|----------|
| DNA extraction | 750 € |
| PCR reactives | 2.100 € |
| Pyrosequencing analysis | 9.000€ |
| Fungible | 950 € |
| SERVICES | |
| Sample transport | 339 € |
| OTHERS | |
| Technical | 4.800 € |
| Overhead IDIBGI (30%) | 5096,7 |
| Total | 23.036 € |